CLINICAL TRIAL: NCT07224373
Title: A Phase 1b, Open-label, Multi-center, Randomized Study Evaluating the Safety and Tolerability of AZD0120, an Autologous CD19/BCMA Targeting Chimeric Antigen Receptor T-cells, in Adults With Refractory Relapsing or Progressive Multiple Sclerosis
Brief Title: An Open-label Study of AZD0120 in Adults With Multiple Sclerosis
Acronym: ZENITH
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D831DC00001; 29707 (Registry Identifier: IND)
Record Dates: First submitted 2025-10-21; First posted 2025-11-04 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: AZD0120; Multiple Sclerosis; MS; RMS; PMS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm/Group 1: AZD0120 RMS (Experimental): AZD0120 RMS
  Interventions: Biological: AZD0120 - Regimen 1; Biological: AZD0120 - Regimen 2
- Arm/Group 2: AZD0120 PMS (Experimental): AZD0120 PMS
  Interventions: Biological: AZD0120 - Regimen 1; Biological: AZD0120 - Regimen 2

INTERVENTIONS:
Biological: AZD0120 - Regimen 1 — Regimen 1, infusion of AZD0120
Biological: AZD0120 - Regimen 2 — Regimen 2, infusion of AZD0120

SUMMARY:
This trial is a Phase 1b, open-label, multi-center, clinical study of AZD0120, a BCMA/CD19 dual targeting CAR+ T-cell therapy, to evaluate the safety and tolerability in adult participants with Multiple Sclerosis.

DETAILED DESCRIPTION:
This study will evaluate AZD0120 for safety, including DLTs and TEAEs, by the SRC for determination of the Recommended Phase 2 dose for each disease cohort. Approximately 9-12 participants will be evaulated per disease cohort.

ELIGIBILITY:
Participants are eligible to be included in the study only if all of the following criteria apply:

Age

1. Age ≥ 18-years-old to ≤ 75-years-old at the time of consent

   Type of Participant and Disease Characteristics
2. Written informed consent in accordance with federal, local, and institutional guidelines
3. Adequate physiological function and reserve at screening

   RMS Cohort Specific Inclusion Criteria
4. Diagnosis of RMS according to the 2017 McDonald Criteria (Thompson et al 2018) or diagnosis of relapsing, active SPMS according to Lublin et al 2014.
5. Participants should have an EDSS of ≤ 6.5 at screening.
6. Evidence of active disease(clinical relapses and MRI activities within 2 years prior to screening), or intolerance, while on a high efficacy disease-modifying therapy for ≥ 6 months.

   PMS Cohort Specific Inclusion Criteria
7. Diagnosis of PPMS according to the 2017 McDonald Criteria (Thompson et al 2018) and/or diagnosis of not active progressive SPMS according to Lublin et al 2014.
8. Participants must have an EDSS of ≥ 3.0 and ≤ 6.5 at screening.
9. Inadequate response ≥ 1 heDMT with ≥ 6 months treatment or intolerance.

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

1. Any prior CAR-T or CAR-NK cell exposure.
2. Underwent splenectomy within 12 months prior to signing the ICF.
3. Received a solid organ transplant at any time or on an active transplant waiting list.
4. Prior treatment with autologous hematopoietic stem cell transplantation or total lymphoid irradiation.
5. Cardiac conditions or any other significant cardiac condition that would present undue risk to the participant in the investigator's opinion:
6. Any other central nervous system disease including epilepsy, convulsive seizures, organic encephalopathy syndrome, non-MS related paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease or associated movement disorder, psychosis, CNS vasculitis, or any other neurological disease that may impact the ability to evaluate neurotoxicity. History of a seizure disorder even if the seizure disorder is well controlled with anti-epileptics.
7. Participant has significant psychiatric condition (active or history of).
8. History of other immune-mediated disease that required continued systemic immunosuppression/systemic disease-modifying agents.
9. Evidence of clinically significant bleeding or active bleeding diathesis within 90 days before screening
10. History of malignancy or ongoing treatment for prior malignancy.
11. Inborn error of immunity and/or primary immunodeficiency.
12. Seropositive for HIV.
13. Active viral (any etiology, HBV, HCV) hepatitis are excluded.
14. Major surgery within 4 weeks prior to apheresis or lymphodepletion or has surgery planned during the study or within 4 weeks after study treatment administration.
15. Pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 1 year after receiving study treatment, whichever is longer.
16. Unwilling or unsafe to proceed with CSF exams based on coagulopathy or anatomy or other considerations in the judgment of the study investigator.
17. Any contraindications to LP.
18. Participants not willing, able, or are unsafe to take MRI scans as per protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2028-12-07 (Estimated); Study Completion 2028-12-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety, and tolerability of AZD0120 in participants with MS (disease cohort 1: RMS; disease cohort 2: PMS) | Day 1 to day 29, and over 104 weeks
  Incidence and severity of Dose Limiting Toxicity (DLT) over 104 weeks following AZD0120 administration.
Evaluate the safety, and tolerability of AZD0120 in participants with MS (disease cohort 1: RMS; disease cohort 2: PMS) | Day 1 to day 29, and over 104 weeks
  Incidence and severity of Adverse Events (AE) over 104 weeks following AZD0120 administration.
Evaluate the safety, and tolerability of AZD0120 in participants with MS (disease cohort 1: RMS; disease cohort 2: PMS) | Day 1 to day 29, and over 104 weeks
  Incidence and severity of Serious Adverse Events (SAE) over 104 weeks following AZD0120 administration.
Evaluate the safety, and tolerability of AZD0120 in participants with MS (disease cohort 1: RMS; disease cohort 2: PMS) | Day 1 to day 29, and over 104 weeks
  Incidence and severity of Treatment Emergent Adverse Events (TEAE) over 104 weeks following AZD0120 administration.

SECONDARY OUTCOMES:
Evaluate the optimum regimen with AZD0120 in MS participants to determine the RP2D in each disease cohort | Over 104 weeks
  Change from baseline in peripheral B-cell counts following AZD0120 administration
Evaluate the optimum regimen with AZD0120 in MS participants to determine the RP2D in each disease cohort | Over 104 weeks
  CK parameters in peripheral B-cell counts following AZD0120 administration
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Annualized Relapse Rate (ARR) over 104 weeks (RMS cohort only)
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Time to onset participants with CDP-12 over 104 weeks
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Proportion of participants with CDP-12 over 104 weeks
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Time to onset participants with CDP-24 over 104 weeks
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Proportion of participants with CDP-24 over 104 weeks
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Proportion of participants achieving CDI
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Change from baseline in 9HPT (9-Hole Peg Test)
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Change from baseline in T25FW (Timed 25-Foot Walk)
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Change from baseline in EDSS (Expanded Disability Status Scale)
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Change from baseline in SDMT (Symbol Digit Modalities Test)
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Proportion of participants with NEDA-3 (No Evidence of Disease Activity)
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Proportion of participants with PIRA (Progression Independent of Relapse Activity)
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Change from screening in MRI parameters including: mean number of Gd+ T1 lesions over time
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Change from screening in MRI parameters including: mean number of new or enlarging T2 hyperintense lesions
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Change from screening in MRI parameters including brain volume
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Change in MRI parameters including: mean number of Gd+ T1 lesions over time.
Evaluate the preliminary efficacy of AZD0120 in RMS and PMS | Over 104 weeks
  Change in MRI parameters including: mean number of new or enlarging T2 hyperintense lesions
Investigate the effects of AZD0120 on the function and quality of life of participants with MS | Over 104 weeks
  Change in SF-36v2 from baseline
Investigate the effects of AZD0120 on the function and quality of life of participants with MS | Over 104 weeks
  Change in Neuro-QoL-fatigue from baseline
Characterize the CK and PD of AZD0120 in participants with MS | Over 104 weeks
  Quantification of CAR transgene levels of AZD0120 in blood and CSF.
Characterize the CK and PD of AZD0120 in participants with MS | Over 104 weeks
  Cmax
Characterize the CK and PD of AZD0120 in participants with MS | Over 104 weeks
  AUC(0-28).
Characterize the CK and PD of AZD0120 in participants with MS | Over 104 weeks
  AUClast.
Characterize the CK and PD of AZD0120 in participants with MS | Over 104 weeks
  Clast.
Characterize the CK and PD of AZD0120 in participants with MS | Over 104 weeks
  Tmax.
Characterize the CK and PD of AZD0120 in participants with MS | Over 104 weeks
  Tlast.
Characterize the CK and PD of AZD0120 in participants with MS | Over 104 weeks
  B-cell counts
To monitor the incidence of vector-derived RCL | Over 104 weeks
  Proportion of participants with detectable RCL at pre-specified post infusion timepoints
To assess the immunogenicity of AZD0120 in participants. | over 104 weeks
  Proportion of participants who develop anti- AZD0120 antibodies
To assess the immunogenicity of AZD0120 in participants. | over 104 weeks
  Time to development of anti-AZD0120 antibodies
To assess the immunogenicity of AZD0120 in participants. | over 104 weeks
  Changes in anti-AZD0120 antibody titers over 104 weeks

CONTACTS AND LOCATIONS:
Locations (12):
- United States (8):
  - Research Site, Tucson, Arizona
  - Research Site, Aurora, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Seattle, Washington
  - Research Site, Milwaukee, Wisconsin
- Australia (3):
  - Research Site, Liverpool
  - Research Site, Melbourne
  - Research Site, Waratah
- Research Site, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No